CLINICAL TRIAL: NCT07365592
Title: A Phase Ib/II Study of Neoadjuvant Chemotherapy Combined With Anti-PD-1 Antibody and DPP4 Inhibitor Sitagliptin for Locally Advanced pMMR Colorectal Cancer
Brief Title: Neoadjuvant Chemotherapy, Anti-PD-1 Antibody and Sitagliptin for Locally Advanced pMMR CRC
Acronym: Neo-CD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jun Li, Chief, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SAHZU Jun LI
Record Dates: First submitted 2025-12-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Capecitabine; spartalizumab; Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Intervention Model Description: Phase Ib Component The study adopts the 3+3 design, with sitagliptin set at three dose groups: 100 mg/day, 200 mg/day, and 400 mg/day.
  Enrollment starts with 3 patients in Group 1. Dose escalates if no DLT; adds 3 patients if 1 DLT occurs. Escalation continues if ≤1/6 have DLT; stops and de-escalates if ≥2/6 have DLT. The study includes 9-18 patients, with no -1 dose group; the lower safe dose becomes MTD if needed.
  Phase II Component The current study presets the TRG 0/1 rate at 20% for the XELOX chemotherapy group. The study expects a TRG 0/1 rate of 30% in the investigational group, representing a 10% relative increase in significant tumor regression compared to standard therapy.
  This is a prospective, multicenter, two-stage randomized controlled interventional study based on a Bayesian adaptive design, with a maximum sample size of 120 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- XELOX+sitagliptin+anti-PD-1 (Experimental): XELOX (oxaliplatin + capecitabine), sitagliptin and PD-1 monoclonal antibody
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Anti-PD-1 monoclonal antibody; Drug: Sitagliptin (DPP4 inhibitor)
- XELOX (Active Comparator): XELOX (oxaliplatin + capecitabine)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 for inducing chemotherapy in Day 1 every 3 weeks and repeat for two cycles.
Drug: Capecitabine — Oral Capecitabine 1000 mg/m2 twice daily combined with oxaliplatin chemotherapy in Day 1 to Day 14 every 3 weeks and repeat for 2 cycles.
Drug: Anti-PD-1 monoclonal antibody — Anti-PD1 antibody 200mg/m2 in Day 1 after oxaliplatin Chemotherapy. Repeat every 3 weeks for 2 cycles.
  Arms: XELOX+sitagliptin+anti-PD-1
Drug: Sitagliptin (DPP4 inhibitor) — Oral sitagliptin twice daily combined with oxaliplatin chemotherapy in Day 1 to Day 14 every 3 weeks and repeat for 2 cycles.
  In the phase Ib study, sitagliptin set at three dose groups: 100 mg/day, 200 mg/day, and 400 mg/day, and the primary endpoint of Ib study is to determine the DLT and recommended phase II dose (RP2D).
  The appropriate dose level of sitagliptin will be set based on the result of Ib study.
  Arms: XELOX+sitagliptin+anti-PD-1

SUMMARY:
This is an open-label, multicenter, phase Ib/II combined trial of sitagliptin, XELOX chemotherapy regimen, and PD-1 monoclonal antibody in the treatment of proficient mismatch repair locally advanced colorectal cancer.

DETAILED DESCRIPTION:
Most colorectal cancer (CRC) cases are classified as proficient mismatch repair (pMMR) CRC. This subtype is insensitive to single-agent immunotherapy, with chemotherapy remaining the primary pharmacotherapeutic intervention. Approximately 30% of colon cancer patients develop recurrence and metastasis following initial radical resection combined with 6 months of adjuvant chemotherapy.

Neoadjuvant chemotherapy (NACT) for tumor downstaging and survival improvement represents a standard approach for locally advanced tumors. However, its application is limited to select rectal cancer populations, and its role in colon cancer remains controversial-primarily due to inadequate tumor regression observed with current regimens. Given that deep tumor regression correlates with improved survival, there is a critical need to enhance NACT efficacy.

Neo-CD adopts a combined phase Ib/II study design. Phase Ib Component

* Design: Single-center trial utilizing the traditional 3+3 dose-escalation principle.
* Objectives:

  1. Evaluate the safety of sitagliptin in combination with XELOX (oxaliplatin + capecitabine) and anti-PD-1 monoclonal antibody as neoadjuvant therapy for CRC.
  2. Determine the recommended phase II dose (RP2D) of sitagliptin.
  3. Explore the combination's potential for significant tumor regression and modulation of the tumor immune microenvironment.

Phase II Component

* Design: Prospective, multicenter, randomized controlled superiority trial.
* Objective: Compare the efficacy of neoadjuvant XELOX + sitagliptin + anti-PD-1 versus standard neoadjuvant XELOX in locally advanced CRC, with a focus on significant tumor regression (TRG 0/1 rate).

Study Procedures All participants will receive 2 cycles of the assigned neoadjuvant treatment, followed by radical surgery.

Primary Endpoints

* Phase Ib: Incidence of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicity (DLT).
* Phase II: Proportion of patients achieving tumor regression grade 0/1 (TRG 0/1).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed colorectal adenocarcinoma
* Age ≥18 years old and ≤75 years old
* MRI/CT stage T3-4aNany and TanyN1-2, without distant metastasis
* Life expectancy of 1 year The above
* Informed consent, no contraindications to chemotherapy exist
* pMMR diagnosed by IHC

Exclusion Criteria:

* Refused to participate in this study
* Multifocal colorectal cancer
* Past history of malignant tumors, except for basal cell carcinoma/papillary thyroid carcinoma/various types of carcinoma in situ
* Unable to receive chemotherapy , such as but not limited to bone marrow suppression, etc
* Major organ diseases (such as but not limited to COPD, coronary heart disease and renal insufficiency, etc.) acute attack and or severe acute infectious diseases (such as but not limited to hepatitis, pneumonia and myocarditis, etc.),
* ASA score> 3
* Mental disorder or illiteracy or language and communication barriers cannot understand the research plan
* Colorectal tumor has obstruction or high risk of obstruction and or there is bleeding and/or perforation
* Peripheral sensory nerve disorder, unable to receive oxaliplatin chemotherapy
* Lateral pelvic lymph node metastasis (mainly supplied by internal iliac artery)
* Pregnancy or breastfeeding
* Unable to accept MRI examination
* Consecutive use of glucocorticoids for more than 3 days within 1 month before signing the consent form
* Diabetes or impaired glucose tolerance who may require drug intervention
* Other scenarios deemed inappropriate by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From date of first chemotherapy until the date of patients were discharged from hospital after receiving radical surgery, up to 20 weeks
  for Ib study
Dose limiting toxicities (DLTs) | The DLT observation period is from the day1 of the first cycle(C1D1) to the start of the day1 of the second cycle(C2D1) dosing, each cycle is 21 days.
  for Ib study
Proportion of patients achieving tumor regression grade 0/1 (TRG 0/1) | 1 day of postoperative pathological examination.
  for II study

SECONDARY OUTCOMES:
Surgical Complication | within 30 days since operation
  for II study
Proportion of patients achieving tumor regression grade 3 (TRG 3) | 1 day of postoperative pathological examination.
  for II study
Adverse events (AEs) | From date of first chemotherapy until the date of patients were discharged from hospital after receiving radical surgery, up to 20 weeks
  for II study
Proportion of patients achieving tumor regression grade 0/1 | 1 day of postoperative pathological examination.
  for Ib study
Proportion of patients achieving pathological Complete Response | 1 day of postoperative pathological examination.
  for Ib study
Proportion of patients achieving Major Pathologic Response | 1 day of postoperative pathological examination.
  for Ib study
Area Under the Curve | From date of first chemotherapy until the date of patients were discharged from hospital after receiving radical surgery, up to 20 weeks
  for Ib study；quantitative measure of the total exposure of the body to a drug over a specific time period.
Maximum Concentration | From date of first chemotherapy until the date of patients were discharged from hospital after receiving radical surgery, up to 20 weeks
  for Ib study; highest plasma or blood concentration of a drug achieved in the body after its administration.
Time to Maximum Concentration | From date of first chemotherapy until the date of patients were discharged from hospital after receiving radical surgery, up to 20 weeks
  for Ib study; the length of time required for a drug to reach its maximum (peak) plasma or blood concentration in the systemic circulation after administration.
Clearance | From date of first chemotherapy until the date of patients were discharged from hospital after receiving radical surgery, up to 20 weeks
  for Ib study; the volume of plasma or blood completely cleared of a drug per unit time by the body's eliminating organs
Half-Life | From date of first chemotherapy until the date of patients were discharged from hospital after receiving radical surgery, up to 20 weeks
  for Ib study; the specific time required for the plasma or blood concentration of a drug in the systemic circulation to decrease by half from its peak level or steady-state level

OTHER OUTCOMES:
DPP4 activity in peripheral blood and tumor tissues | From date of first chemotherapy until the date of patients were discharged from hospital after receiving radical surgery, up to 20 weeks
  for Ib study;
The changes in the immunoprofile of the tumor tissue sample among TRG0/1 and TRG2/3 patients | 3 months after surgery
  By using single-cell analysis, we comprehensively characterized the immune landscape in the tumor sample of CRC patients before and after neoadjuvant treatment.
2-year overall survival | 2-year after surgery
  for II study; The proportion of all study cases in which no death from any cause occurred within 2 years after surgery
2-year Disease-free survival | From date of first chemotherapy until the date of first documented recurrence of tumor or date of death from any cause，whichever came first，assessed up to 24 months.
  From date of first chemotherapy until the date of first documented recurrence of tumor or date of death from any cause，whichever came first，assessed up to 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided